CLINICAL TRIAL: NCT00078819
Title: Placebo-controlled Multicenter Study With Etanercept to Determine Safety and Efficacy in Pediatric Subjects With Plaque Psoriasis (PEDS)
Brief Title: Etanercept (Enbrel®) in Psoriasis - Pediatrics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20030211
Record Dates: First submitted 2004-03-05; First posted 2004-03-09 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-05

CONDITIONS: Psoriasis
Keywords: Pediatric Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12). Participants with a > 50% worsening (ie, increase) in Psoriasis Area and Severity Index (PASI) score at or after week 4 compared with baseline and an increase of at least 4 points at 1 visit, or an increase of more than 25% and by a minimum of 4 points at each of two consecutive visits, could escape to etanercept 0.8 mg/kg once a week up to week 12.
  Participants received open-label etanercept 0.8 mg/kg once a week during the 24-week, open-label treatment period (weeks 13 to 36).
  At week 36, participants with PASI 50 at week 24 or PASI 75 at week 36 were re-randomized to placebo or etanercept in the 12-week double-blind, withdrawal-retreatment period (weeks 37 to 48).
  Interventions: Drug: Placebo
- Etanercept (Experimental): Participants received 0.8 mg/kg etanercept administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12). Participants with a > 50% worsening (ie, increase) in Psoriasis Area and Severity Index (PASI) score at or after week 4 compared with baseline and an increase of at least 4 points at 1 visit, or an increase of more than 25% and by a minimum of 4 points at each of two consecutive visits, could escape to etanercept 0.8 mg/kg once a week up to week 12.
  Participants received open-label etanercept 0.8 mg/kg once a week during the 24-week, open-label treatment period (weeks 13 to 36).
  At week 36, participants with PASI 50 at week 24 or PASI 75 at week 36 were re-randomized to placebo or etanercept in the 12-week double-blind, withdrawal-retreatment period (weeks 37 to 48).
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept 0.8 mg/kg (up to an intended dose of 50 mg) by subcutaneous injection once a week
  Other Names: Enbrel®
  Arms: Etanercept
Drug: Placebo — Placebo matching to etanercept administered by subcutaneous injection once a week
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of etanercept (Enbrel®) in children with Psoriasis.

DETAILED DESCRIPTION:
On enrollment, participants underwent randomization in a 1:1 ratio to receive placebo or etanercept during the initial double-blind period. Participants could enter an escape group and receive open-label etanercept until week 12 if, at or after week 4, their Psoriasis Area and Severity Index (PASI) score either increased by more than 50% over baseline and by a minimum of 4 points at one visit or increased by more than 25% and by a minimum of 4 points at each of two consecutive visits.

During the open-label treatment period, all patients (including those who entered the escape group) received open-label etanercept. Participants who did not achieve PASI 50 at week 24 or PASI 75 at week 36 could discontinue the study or add topical standard-of-care therapy (low-to-moderate-potency topical corticosteroids) and continue to receive open-label etanercept until week 48.

At week 36, participants with PASI 50 at week 24 or PASI 75 at week 36 were randomly assigned to placebo or etanercept for 12 weeks in the withdrawal period. Participants in whom PASI 75 was lost resumed open-label etanercept through week 48 in the re-treatment period.

ELIGIBILITY:
* Patients with plaque psoriasis
* Patient may not receive certain psoriasis medications during the study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2004-09-08 (Actual); Primary Completion 2006-02-01 (Actual); Study Completion 2007-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Langley RG, Kasichayanula S, Trivedi M, Aras GA, Kaliyaperumal A, Yuraszeck T, Gibbs J, Gibbs M, Kricorian G, Paller AS. Pharmacokinetics, Immunogenicity, and Efficacy of Etanercept in Pediatric Patients With Moderate to Severe Plaque Psoriasis. J Clin Pharmacol. 2018 Mar;58(3):340-346. doi: 10.1002/jcph.1029. Epub 2017 Nov 6. PMID 29106714
- [Background] Landells I, Paller AS, Pariser D, Kricorian G, Foehl J, Molta C, Freundlich B. Efficacy and safety of etanercept in children and adolescents aged > or = 8 years with severe plaque psoriasis. Eur J Dermatol. 2010 May-Jun;20(3):323-8. doi: 10.1684/ejd.2010.0911. Epub 2010 Feb 25. PMID 20185386
- [Background] Langley RG, Paller AS, Hebert AA, Creamer K, Weng HH, Jahreis A, Globe D, Patel V, Orlow SJ. Patient-reported outcomes in pediatric patients with psoriasis undergoing etanercept treatment: 12-week results from a phase III randomized controlled trial. J Am Acad Dermatol. 2011 Jan;64(1):64-70. doi: 10.1016/j.jaad.2010.02.060. Epub 2010 Jul 8. PMID 20619489
- [Background] Paller AS, Eichenfield LF, Langley RG, Leonardi CL, Siegfried EC, Creamer K, Kricorian G. Subgroup analyses of etanercept in pediatric patients with psoriasis. J Am Acad Dermatol. 2010 Aug;63(2):e38-41. doi: 10.1016/j.jaad.2009.11.001. No abstract available. PMID 20633781
- [Background] Paller AS, Siegfried EC, Langley RG, Gottlieb AB, Pariser D, Landells I, Hebert AA, Eichenfield LF, Patel V, Creamer K, Jahreis A; Etanercept Pediatric Psoriasis Study Group. Etanercept treatment for children and adolescents with plaque psoriasis. N Engl J Med. 2008 Jan 17;358(3):241-51. doi: 10.1056/NEJMoa066886. PMID 18199863
- [Background] Siegfried EC, Eichenfield LF, Paller AS, Pariser D, Creamer K, Kricorian G. Intermittent etanercept therapy in pediatric patients with psoriasis. J Am Acad Dermatol. 2010 Nov;63(5):769-74. doi: 10.1016/j.jaad.2009.10.046. Epub 2010 Sep 15. PMID 20833444
- [Background] Varni JW, Globe DR, Gandra SR, Harrison DJ, Hooper M, Baumgartner S. Health-related quality of life of pediatric patients with moderate to severe plaque psoriasis: comparisons to four common chronic diseases. Eur J Pediatr. 2012 Mar;171(3):485-92. doi: 10.1007/s00431-011-1587-2. Epub 2011 Sep 30. PMID 21960290
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20030211.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This 48-week study was conducted at 42 sites in the United States and Canada. The first participant was enrolled on September 8, 2004, and the last participant on November 29, 2005.
Pre-assignment Details: On enrollment, participants underwent randomization at a 1:1 ratio by an interactive voice-response system.
Groups:
- Placebo: Participants randomized to receive placebo administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12). Participants with a > 50% worsening (ie, increase) in Psoriasis Area and Severity Index (PASI) score at or after week 4 compared with baseline and an increase of at least 4 points at 1 visit, or with an increase of more than 25% and by a minimum of 4 points at each of two consecutive visits, could escape to etanercept 0.8 mg/kg once a week up to week 12.
  Participants (including those who escaped to etanercept) received open-label etanercept 0.8 mg/kg once a week during the 24-week, open-label treatment period (weeks 13 to 36).
  Participants who did not achieve PASI 50 at week 24 or PASI 75 at week 36 (incomplete response) could discontinue the study or continue to receive open-label etanercept with a topical standard-of-care until week 48.
- Etanercept: Participants randomized to receive 0.8 mg/kg etanercept administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12). Participants with a more than 50% worsening (ie, increase) in PASI score at or after week 4 compared with baseline and an increase of at least 4 points at 1 visit, or with an increase of more than 25% and by a minimum of 4 points at each of two consecutive visits, could escape to etanercept 0.8 mg/kg once a week up to week 12.
  Participants (including those who escaped to etanercept) received open-label etanercept 0.8 mg/kg once a week during the 24-week, open-label treatment period (weeks 13 to 36).
  Participants who did not achieve PASI 50 at week 24 or PASI 75 at week 36 (incomplete response) could discontinue the study or continue to receive open-label etanercept with a topical standard-of-care until week 48.
- Withdrawal/Re-treatment Period: Placebo: At week 36, participants with a PASI 75 response were re-randomized to receive placebo once a week for 12-weeks in the double-blind withdrawal period (weeks 37 to 48).
  Participants who relapsed (defined as a loss of PASI 75 response) were to resume open-label treatment with 0.8 mg/kg etanercept once a week until week 48 (re-treatment period).
- Withdrawal/Re-treatment Period: Etanercept: At week 36, participants with a PASI 75 response were re-randomized to receive 0.8 mg/kg etanercept once a week for 12-weeks in the double-blind, withdrawal period (weeks 37 to 48).
  Participants who relapsed (defined as a loss of PASI 75 response) were to resume open-label treatment with 0.8 mg/kg etanercept once a week until week 48 (re-treatment period).
Period: Double-blind Treatment Period: Week 1-12
Arm/Group | Placebo | Etanercept | Withdrawal/Re-treatment Period: Placebo | Withdrawal/Re-treatment Period: Etanercept
Started | 105 | 106 | 0 | 0
Entered Escape | 27 | 5 | 0 | 0
Completed (Includes participants who escaped early) | 104 | 105 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Open-label Treatment Period: Weeks 13-36
Arm/Group | Placebo | Etanercept | Withdrawal/Re-treatment Period: Placebo | Withdrawal/Re-treatment Period: Etanercept
Started | 103 (One participant discontinued before starting the open-label period) | 105 | 0 | 0
Completed (Includes participants who completed week 36 with a PASI response) | 63 | 75 | 0 | 0
Not Completed | 40 | 30 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Not completed — Incomplete Responders | 34 | 25 | 0 | 0
Period: Withdrawal Period: Weeks 37-48
Arm/Group | Placebo | Etanercept | Withdrawal/Re-treatment Period: Placebo | Withdrawal/Re-treatment Period: Etanercept
Started | 0 | 0 | 69 (Participants who completed week 36 with a PASI response) | 69 (Participants who completed week 36 with a PASI response)
Received Study Drug | 0 | 0 | 69 | 68
Completed | 0 | 0 | 40 (Defined as continuing to receive blinded study drug through week 48) | 55 (Defined as continuing to receive blinded study drug through week 48)
Not Completed | 0 | 0 | 29 | 14
Not completed — Entered Retreatment | 0 | 0 | 29 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Period: Re-treatment Period
Arm/Group | Placebo | Etanercept | Withdrawal/Re-treatment Period: Placebo | Withdrawal/Re-treatment Period: Etanercept
Started | 0 | 0 | 29 | 13
Received Study Drug | 0 | 0 | 30 (One additional participant received re-treatment without having disease relapse) | 12
Completed | 0 | 0 | 29 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants randomized to receive placebo administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12).
- Etanercept: Participants randomized to receive 0.8 mg/kg etanercept administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12).
- Total: Total of all reporting groups
Arm/Group | Placebo | Etanercept | Total
Number analyzed (Participants) | 105 | 106 | 211
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 13.00 [4.0 to 17.0] | 14.00 [4.0 to 17.0] | 13.00 [4.0 to 17.0]
Age, Customized [Count of Participants; unit: Participants]
  4 to 11 years | 38 | 38 | 76
  12 to 17 years | 67 | 68 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 103
  Male | 53 | 55 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 75 | 83 | 158
  Black or African American | 8 | 3 | 11
  Hispanic or Latino | 14 | 8 | 22
  Asian | 6 | 9 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 2 | 2 | 4
Duration of Psoriasis [Median (Full Range); unit: years] | 5.80 [0.3 to 15.8] | 6.80 [0.3 to 17.9] | 5.90 [0.3 to 17.9]
Psoriasis Area and Severity Index (PASI) [Median (Full Range); unit: units on a scale] — The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by erythema (reddening), induration (plaque thickness) and desquamation (scaling) scored on a scale from 0 (none) to 4 (very severe), together with the percentage of the area affected, rated on a scale from 0 (no involvement) to 6 (90% to 100% involvement). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
  units on a scale | 16.40 [12.0 to 56.7] | 16.70 [12.0 to 51.6] | 16.40 [12.0 to 56.7]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a ≥ 75% Improvement in Psoriasis Area and Severity Index Score (PASI 75) at Week 12
Description: The percentage of participants who achieved 75% or greater improvement (decrease) from baseline in PASI score after 12 weeks of treatment. The PASI score is a combination of the intensity of psoriasis, assessed by erythema (reddening), induration (plaque thickness) and desquamation (scaling) scored on a scale from 0 (none) to 4 (very severe), together with the percentage of the area affected, rated on a scale from 0 (no involvement) to 6 (90% to 100% involvement). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
  Participants who entered the escape arm or had missing data at week 12 were considered non-responders.
Time Frame: Baseline and week 12
Population: The intent-to-treat population included all randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants randomized to receive placebo administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12). Participants with a > 50% worsening (ie, increase) in Psoriasis Area and Severity Index (PASI) score at or after week 4 compared with baseline and an increase of at least 4 points at 1 visit, or with an increase of more than 25% and by a minimum of 4 points at each of two consecutive visits, could escape to etanercept 0.8 mg/kg once a week up to week 12.
- Etanercept: Participants randomized to receive 0.8 mg/kg etanercept administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12). Participants with a more than 50% worsening (ie, increase) in PASI score at or after week 4 compared with baseline and an increase of at least 4 points at 1 visit, or with an increase of more than 25% and by a minimum of 4 points at each of two consecutive visits, could escape to etanercept 0.8 mg/kg once a week up to week 12.
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 105 | 106
percentage of participants | 11.0 | 57.0
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Test type: Superiority — The significance levels for primary and secondary efficacy end points were controlled at 0.05 with the use of a sequential testing scheme in this order: PASI 75, PASI 50, a physician's global assessment of clear or almost clear, percentage improvement from baseline in CDLQI, and PASI 90; p < 0.0001, Cochran-Mantel-Haenszel; Two-sided Cochran-Mantel-Haenszel test stratified by age group

2. Secondary Outcome: Percentage of Participants Achieving a ≥ 50% Improvement in PASI Score (PASI 50) at Week 12
Description: The percentage of participants who achieved 50% or greater improvement from baseline in PASI score after 12 weeks of treatment. PASI is a combination of the intensity of psoriasis, assessed by erythema (reddening), induration (plaque thickness) and desquamation (scaling) scored on a scale from 0 (none) to 4 (very severe), together with the percentage of the area affected, rated on a scale from 0 (no involvement) to 6 (90% to 100% involvement). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
  Participants who entered the escape arm or had missing data at week 12 were considered non-responders.
Time Frame: Baseline and week 12
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 105 | 106
percentage of participants | 23 | 75
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Two-sided Cochran-Mantel-Haenszel test stratified by age group

3. Secondary Outcome: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of Clear (0) or Almost Clear (1) at Week 12
Description: The sPGA is a static measurement based on induration, erythema, and scaling. The sPGA is assessed on a scale from 0 to 5:
  0 = clear (no evidence of plaque elevation, erythema or scaling)
  1. = almost clear (minimal plaque elevation, erythema or scaling)
  2. = mild (mild plaque elevation or scaling, light red coloration)
  3. = moderate (moderate plaque elevation, scaling, light red coloration)
  4. = marked (marked plaque elevation, thick, non-tenacious scale predominates, bright red coloration)
  5. = severe (severe plaque elevation, very thick tenacious scaling, dusky to deep red coloration).
  Participants who entered the escape arm or had missing data at week 12 were considered non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 105 | 106
percentage of participants | 13 | 53
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Two-sided Cochran-Mantel-Haenszel test stratified by age group

4. Secondary Outcome: Percent Improvement From Baseline in Children's Dermatology Life Quality Index (CDLQI) at Week 12
Description: The Children's Dermatology Life Quality Index (CDLQI) was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (Not at all) to 3 (Very much). The total score ranges from 0 to 30, with lower scores indicating better quality of life. If participants were ≥ 13 years old, the text instrument was completed by the participants themselves. Participants ≥ 8 but < 13 years old used the cartoon version of the instrument and participants ≤ 7 years old used the cartoon version of the instrument completed with help from the parents or caregivers.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline Value * 100.
  Participants who entered the escape arm or who had missing data at week 12 were considered to have 0% improvement from baseline.
Time Frame: Baseline and week 12
Population: Intent-to-treat population with available CDLQI data at baseline
Measure: Mean (Standard Error); unit: percent improvement
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 102 | 100
percent improvement | 17.5 (8.3) | 52.3 (6.1)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Van Elteren test; Two-sided van Elteren's test stratified by age group

5. Secondary Outcome: Percentage of Participants Achieving a ≥ 90% Improvement in PASI Score (PASI 90) at Week 12
Description: The percentage of participants who achieved 90% or greater improvement from baseline in PASI score after 12 weeks of treatment. The PASI score is a combination of the intensity of psoriasis, assessed by erythema (reddening), induration (plaque thickness) and desquamation (scaling) scored on a scale from 0 (none) to 4 (very severe), together with the percentage of the area affected, rated on a scale from 0 (no involvement) to 6 (90% to 100% involvement). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
  Participants who entered the escape arm or had missing data at week 12 were considered non-responders.
Time Frame: Baseline and week 12
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 105 | 106
percentage of participants | 7 | 27
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Two-sided Cochran-Mantel-Haenszel test stratified by age group

6. Secondary Outcome: Number of Participants With Adverse Events During the Double-blind Treatment Period
Description: The severity assessment for adverse events and infections was done using the Common Toxicity Criteria (CTC) Version 2.0, where Grade 0 = no toxicity, Grade 1 = mild toxicity, Grade 2 = moderate toxicity, Grade 3 = severe toxicity, Grade 4 = life-threatening toxicity.
  Serious adverse events were any events that suggested a significant hazard or side effect, regardless of the investigator's or sponsor's opinion on the relationship to study medication. These included, but were not limited to, events at any dose that were fatal, life threatening, required in-patient hospitalization or prolonged hospitalization, were a persistent or significant disability/incapacity, or were a congenital abnormality/birth defect. Medical events that jeopardized a participant, required intervention to prevent one of the above outcomes, or resulted in urgent investigation could be considered serious.
Time Frame: 12 weeks
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants randomized to receive placebo administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12). Adverse events are reported up until escape for participants who escaped to etanercept.
- Etanercept: Participants randomized to receive 0.8 mg/kg etanercept administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12).
  Adverse events are reported up until escape for participants who escaped to etanercept.
- Escape: Etanercept: Participants with a > 50% worsening (ie, increase) in PASI score at or after week 4 compared with baseline and an increase of at least 4 points at 1 visit, or with an increase of more than 25% and by a minimum of 4 points at each of two consecutive visits, escaped to etanercept 0.8 mg/kg once a week up to week 12.
Arm/Group | Placebo | Etanercept | Escape: Etanercept
Number analyzed (Participants) | 105 | 106 | 32
Participants
  Any adverse event | 62 | 68 | 16
  Non-infectious adverse event | 46 | 42 | 9
  Infection | 33 | 50 | 9
  Serious non-infectious adverse event | 0 | 0 | 0
  Serious infection | 0 | 0 | 0
  Death | 0 | 0 | 0
  Grade 3 non-infectious adverse event | 3 | 0 | 0
  Grade 3 infection | 0 | 0 | 0
  Non-infectious AE leading to withdrawal from Study | 0 | 1 | 0
  Infection leading to withdrawal from Study | 0 | 0 | 0
  Injection site reaction | 5 | 7 | 1

7. Secondary Outcome: Etanercept Serum Concentration
Description: Serum concentrations for etanercept were measured by using a validated enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) was 0.627 ng/mL.
Time Frame: Day 1 (predose), week 12, week 24, and week 48
Population: Participants assigned to etanercept at any time during the study, with available data.
  Week 12 excludes participants assigned to placebo who escaped to etanercept. Week 48 includes participants randomized to etanercept at week 36 and remaining on etanercept to week 48. Participants randomized to placebo and retreated with etanercept are excluded.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Etanercept
Number analyzed (Participants) | 208
ng/mL
  Day 1: number analyzed (Participants) | 124
  Day 1 | 1.50 (3.13)
  Week 12: number analyzed (Participants) | 99
  Week 12 | 1614 (828)
  Week 24: number analyzed (Participants) | 191
  Week 24 | 2104 (1255)
  Week 48: number analyzed (Participants) | 106
  Week 48 | 1650 (1126)

ADVERSE EVENTS:
Time Frame: Double-blind treatment period: 12 weeks Escape to etanercept: from time of escape to week 12 (maximum of 8 weeks) Open-label treatment period: 24 weeks Incomplete response: From date of incomplete response to week 48 (maximum of 24 weeks) Withdrawal Period: 12 weeks Re-treatment Period: From date of re-treatment to week 48 (maximum of 8 weeks)
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Double-blind Period: Placebo: Participants received placebo administered by subcutaneous injection once a week during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12).
- Double-blind Period: Etanercept 0.8 mg/kg QW: Participants received 0.8 mg/kg etanercept administered by subcutaneous injection once a week (QW) during the 12-week, double-blind, placebo-controlled treatment period (day 1 to week 12).
- Double-blind Period: Escape to Etanercept 0.8 mg/kg QW: Participants with a > 50% worsening (ie, increase) in PASI score at or after week 4 compared with baseline and an increase of at least 4 points at 1 visit, or with an increase of more than 25% and by a minimum of 4 points at each of two consecutive visits, escaped to etanercept 0.8 mg/kg once a week up to week 12.
- Open-label Period: Etanercept 0.8 mg/kg QW: Participants received open-label etanercept 0.8 mg/kg once a week during the 24-week, open-label treatment period (weeks 13 to 36).
- Open-label Period Incomplete Response: Etanercept 0.8 mg/kg QW: Participants who did not achieve PASI 50 at week 24 or PASI 75 at week 36 continued to receive open-label etanercept 0.8 mg/kg QW plus optional topical standard-of-care therapy (low-to-moderate-potency topical corticosteroids) until week 48.
- Withdrawal Period: Placebo: At week 36, participants with a PASI 75 response were re-randomized to receive placebo once a week for 12 weeks in the double-blind, withdrawal period (weeks 37 to 48) or until relapse (loss of PASI 75 response).
- Withdrawal Period: Etanercept 0.8 mg/kg QW: At week 36, participants with a PASI 75 response were re-randomized to receive 0.8 mg/kg etanercept once a week for 12-weeks in the double-blind, withdrawal period (weeks 37 to 48) or until relapse (loss of PASI 75 response).
- Re-treatment Period: Placebo/Etanercept 0.8 mg/kg QW: Participants randomized to placebo at week 36 who relapsed (loss of PASI 75 response) resumed open-label treatment with 0.8 mg/kg etanercept once a week until week 48.
- Re-treatment Period: Etanercept / Etanercept 0.8 mg/kg QW: Participants randomized to etanercept at week 36 who relapsed (loss of PASI 75 response) resumed open-label treatment with 0.8 mg/kg etanercept once a week until week 48.
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Etanercept 0.8 mg/kg QW | Double-blind Period: Escape to Etanercept 0.8 mg/kg QW | Open-label Period: Etanercept 0.8 mg/kg QW | Open-label Period Incomplete Response: Etanercept 0.8 mg/kg QW | Withdrawal Period: Placebo | Withdrawal Period: Etanercept 0.8 mg/kg QW | Re-treatment Period: Placebo/Etanercept 0.8 mg/kg QW | Re-treatment Period: Etanercept / Etanercept 0.8 mg/kg QW
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/106 | 0/32 | 0/208 | 0/59 | 0/69 | 0/68 | 0/30 | 0/12
Other Adverse Events (participants affected / at risk) | 44/105 | 59/106 | 10/32 | 174/208 | 54/59 | 23/69 | 26/68 | 9/30 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Period: Placebo (N=105) | Double-blind Period: Etanercept 0.8 mg/kg QW (N=106) | Double-blind Period: Escape to Etanercept 0.8 mg/kg QW (N=32) | Open-label Period: Etanercept 0.8 mg/kg QW (N=208) | Open-label Period Incomplete Response: Etanercept 0.8 mg/kg QW (N=59) | Withdrawal Period: Placebo (N=69) | Withdrawal Period: Etanercept 0.8 mg/kg QW (N=68) | Re-treatment Period: Placebo/Etanercept 0.8 mg/kg QW (N=30) | Re-treatment Period: Etanercept / Etanercept 0.8 mg/kg QW (N=12)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 3 | 0 | 11 | 2 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0 | 9 | 4 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 0 | 13 | 3 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4 | 0 | 15 | 6 | 1 | 2 | 0 | 1
Injection Site Bruising (General disorders) | 4 | 1 | 0 | 12 | 3 | 0 | 1 | 0 | 0
Injection Site Pain (General disorders) | 0 | 2 | 0 | 6 | 3 | 0 | 0 | 0 | 1
Injection Site Reaction (General disorders) | 0 | 2 | 0 | 7 | 3 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 12 | 1 | 2 | 2 | 0 | 0
Seasonal Allergy (Immune system disorders) | 1 | 1 | 0 | 4 | 1 | 0 | 0 | 0 | 1
Body Tinea (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1
Conjunctivitis Viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ear Infection (Infections and infestations) | 1 | 2 | 0 | 9 | 2 | 1 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 6 | 3 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 6 | 1 | 13 | 4 | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 3 | 2 | 0 | 13 | 5 | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 8 | 0 | 23 | 2 | 2 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 9 | 8 | 0 | 39 | 12 | 2 | 7 | 0 | 0
Otitis Media (Infections and infestations) | 2 | 0 | 0 | 10 | 5 | 0 | 2 | 1 | 0
Pharyngitis (Infections and infestations) | 4 | 2 | 0 | 13 | 5 | 0 | 0 | 0 | 0
Pharyngitis Streptococcal (Infections and infestations) | 1 | 3 | 1 | 17 | 6 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 12 | 3 | 0 | 2 | 2 | 1
Skin Infection (Infections and infestations) | 1 | 1 | 1 | 8 | 4 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 18 | 4 | 64 | 25 | 7 | 2 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 10 | 4 | 0 | 0 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 13 | 3 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 5 | 0 | 8 | 3 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 13 | 14 | 1 | 42 | 12 | 2 | 6 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 19 | 4 | 5 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 17 | 3 | 2 | 0 | 2 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1 | 20 | 9 | 3 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 9 | 5 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 10 | 4 | 0 | 2 | 0 | 0
Guttate Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 4 | 3 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 5 | 3 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.